CLINICAL TRIAL: NCT04019080
Title: Real-Life Use of Anti-fibrotic Drugs in Patients With Idiopathic Pulmonary Fibrosis in Sweden
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Skold, Professor, Senior consultant, Karolinska University Hospital
Other Study IDs: 180293
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Anti-fibrostic drugs — The real-Life use of anti-fibrotic drugs in patients with idiopathic pulmonary fibrosis in Sweden

SUMMARY:
The objective of the current research project is, by using high quality Swedish registry data, to evaluate use, tolerance and effect of anti-fibrotic drugs in IPF-patients. Secondary study objectives are to determine the clinical profile, determinants of treatment adherence, long-term safety and to describe the patient journey from the first sign of disease to end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* All subjects included in the Swedish IPF-registry

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with idiopathic pulmonary fibrosis included in the Swedish IPF-registry
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Anti-fibrotic drugs among the patients recorded in the Swedish IPF-registry | 2014-2020
  The use of anti-fibrostic drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden